CLINICAL TRIAL: NCT05878782
Title: Occupational Engagement in Alder Adults With Cancer - the Impact of Occupational Therapy (OCEAN-OT): a Multicenter Randomized Controlled Trial
Brief Title: the Impact of Occupational Therapy : a Multicenter Randomized Controlled Trial
Acronym: OCEAN-OT
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: APHP230405
Record Dates: First submitted 2023-05-19; First posted 2023-05-26 (Actual); Last update posted 2023-05-26 (Actual); Status verified 2023-05

CONDITIONS: Elderly Patient; Cancer; Quality of Life
MeSH Terms: conditions — Neoplasms | interventions — Methods

STUDY DESIGN:
Intervention Model Description: A randomized, controlled, superiority trial in 3 parallel arms
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Occupational therapy intervention associated with MCRO assesment. (Experimental): the experimental care of this group will combine the assessment of occupational problems (MCRO) and an occupational therapy intervention.
  Interventions: Other: MCRO+Occupational therapy
- MCRO assessment without intervention (Experimental): This experimental group will have only the MCRO assessment because the occupational problems assessment alone (without intervention) could improve quality of life and occupational performance outcomes, according to the Nielsen, 2019 study
  Interventions: Other: MCRO without intervention
- Usual care (No Intervention): this group will have the usual cancer management care combining specific treatments and supportive care.

INTERVENTIONS:
Other: MCRO+Occupational therapy — Experimental group A will combine the assessment of occupational problems (MCRO) and an occupational therapy intervention.
  Other Names: experimental arm A :Occupational therapy intervention associated with MCRO assesment
  Arms: Occupational therapy intervention associated with MCRO assesment.
Other: MCRO without intervention — Experimental group B will have only the MCRO assessment because the occupational problems assessment alone (without intervention) could improve quality of life and occupational performance outcomes, according to the Nielsen, 2019 study
  Other Names: experimental arm B: MCRO assessment only
  Arms: MCRO assessment without intervention

SUMMARY:
The purpose of this randomized controlled superiority trial is to evaluate the impact of occupational therapy assessment and intervention on the quality of life of elderly cancer patients.

Patients will be randomized into 3 parallel, multicenter arms with patient-reported outcome and blinded evaluator.

* Experimental group A will combine the assessment of occupational problems (MCRO) and an occupational therapy intervention.
* Experimental group B will have only the MCRO assessment because the occupational problems assessment alone (without intervention) could improve quality of life and occupational performance outcomes, according to the Nielsen, 2019 study
* Group C will have the usual cancer management care combining specific treatments and supportive care.

DETAILED DESCRIPTION:
in order to limit the potential grading bias associated with the open-label design, the reassessment at 3 and 6 months will be performed by a different occupational therapist than the one who performed the initial assessment and occupational therapy intervention. For this reason, at least two occupational therapists per geographic area of the centers that include the patients will be included in the project.

ELIGIBILITY:
Inclusion Criteria:

* ≥ 70 years;
* Colorectal, breast, prostate or lung cancer;
* Between 1 and 3 months after the start of cancer treatment depending on the type of treatment (Surgery and/or systemic treatment and/or radiotherapy);
* For curative purposes;
* Affiliated to a social security scheme;
* Living at home;
* Agreeing to participate in the research and having given a free, informed and signed consent

Exclusion Criteria:

* person caring for a patient meeting the above criteria;
* Living with the patient;
* Agreeing to participate in the research and having given free, informed and signed consent

Min Age: 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 232 (Estimated)
Dates: Start 2023-09-01 (Estimated); Primary Completion 2026-05-01 (Estimated); Study Completion 2026-05-01 (Estimated)

PRIMARY OUTCOMES:
Quality of life (QLQ-C30 questionnaire) | 3 months
  Evolution of the EORTC QLQ-C30 role functioning score at 3 months

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Engels C, Marliac Schweitzer S, Blond O, Boulahssass R, David C, Faure H, Gaborit C, Kirscher S, Doyle Lyons K, Machado Antunes L, Morisset L, Pergolotti M, Pierro M, Pineau-Ribas C, Thamie S, Rollot-Trad F, Canoui-Poitrine F. Effects of occupational therapy on quality of life, occupational performance, and occupational satisfaction in older adults with cancer: a multicentre, pragmatic, randomized, controlled trial protocol (OCEAN-OT). BMC Geriatr. 2025 Nov 27;25(1):1064. doi: 10.1186/s12877-025-06535-y. PMID 41310492